CLINICAL TRIAL: NCT02979782
Title: Neurological Outcome After Minimal Invasive Coronary Artery Bypass Graft: a Single-centre Prospective Cohort Study
Brief Title: Neurological Outcome After Minimal Invasive Coronary Artery Bypass Graft
Acronym: NOMICS
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Principal Investigator, Stessel Björn, MD, Jessa Hospital
Other Study IDs: 16.115/anesth16.01
Record Dates: First submitted 2016-11-23; First posted 2016-12-02 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Cognitive Dysfunction; Cerebrovascular Accident; Delirium
Keywords: cardiac surgery; neurological outcome; minimal invasive coronary artery bypass graft (Endo-CABG)
MeSH Terms: conditions — Postoperative Cognitive Complications; Stroke; Delirium | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Endo-CABG, surgical group: the minimal invasive cardiac surgery group
  Interventions: Procedure: Endo-CABG
- PCI, comparative surgical group: a comparative minimal invasive procedure
  Interventions: Procedure: PCI
- Healthy volunteer, control group: to exclude any learning effect or natural variation in neurological testing

INTERVENTIONS:
Procedure: Endo-CABG — minimal invasive cardiac intervention
  Other Names: minimal invasive Coronary Artery Bypass Grafting
  Groups: Endo-CABG, surgical group
Procedure: PCI — stenting procedure
  Other Names: percutaneous coronary intervention
  Groups: PCI, comparative surgical group

SUMMARY:
Primary objectives:

Assessment of the incidence of postoperative cognitive dysfunction (POCD), cerebrovascular accident (CVA), and delirium after minimal invasive coronary artery bypass grafting (Endo-CABG).

Secondary objectives:

* Quality of life, three months after endo-CABG
* Patient satisfaction with endo-CABG and the tests performed
* The influence of various demographic and peri-operative variables on neurological outcome after endo-CABG
* Incidence of fear and depression, 3 months after endo-CABG

DETAILED DESCRIPTION:
Introduction:

Major improvements in surgical techniques, perfusion systems, and perioperative policies have led to improved quality of life of the patient, lower hospitalisation costs, and lower mortality rates in the field of cardiac surgery. However, despite these improvements and improved postoperative care, the neurological outcome after cardiac surgery remains a recurrent issue of interest. The most common neurological disorders after cardiac surgery are postoperative cognitive dysfunction (POCD), cerebrovascular accident (CVA), and delirium. After conventional cardiac surgery (invasive sternotomy procedure) the incidence of these neurological disorders is well studied. POCD has an incidence of 25-50%, CVA has an incidence of 1-5% and delirium has an incidence of 5-15%. These numbers prove that neurological outcome still is a major problem after cardiac surgery.

Postoperative cognitive dysfunction (POCD) is the most common neurological disorder after cardiac surgery. POCD is defined as a disturbance of the brain function, which is causally related to surgery. Due to the multifactorial nature of POCD it is difficult to pinpoint one major cause. testing of POCD is not standardised and is based on the '1995 statement of concensus on assessment of neurobehavioural outcomes after cardiac surgery'. This consensus statement describes the most reliable tests and study design to study POCD in clinical studies.

A battery of tests is described in the consensus statement:

* Rey auditory verbal learning test for verbal memory
* Trailmaking A and B for attention
* Grooved pegboard test for fine motor function

In this study, two additional tests will be performed to assess POCD:

the digit span test to test the short term verbal memory. the digit symbol-coding test to test the processing speed and memory of the patient.

Additional recommendations of the consensus statement to conduct reliable POCD testing are:

* Baseline testing
* At least on assessment of POCD three months postoperatively
* A control group and a comparative group
* The same person tests both pre- and postoperatively
* a clinical neurological investigation is necessary

Cerebrovascular accident (CVA or stroke) is caused by disturbances of the brain blood supply. The main causes of these disturbances are clotted vessels, hypoperfusion, or ruptured vessels in the brain. The risk of CVA is high in the first few days after cardiac surgery. CVA is diagnosed based on neurological evaluation and signs on CT or MRI scan.

Delirium is characterised by attention disorders and fluctuating changes in the mental state of the patient. Delirium is mainly related to surgery and can be diagnosed with the CAM-ICU (confusion assessment method for the intensive care unit).

These neurological complications have a negative effect on the quality of life, healthcare costs and mortality rate after cardiac surgery.

Recently, new developments in cardiac surgery hav led to the introduction of minimal invasive cardiac procedures into practice. These minimal invasive cardiac procedures are proven to be beneficial for the patient. Neurological outcome after minimal invasive cardiac surgery however, is not well studied.

Therefore, the main goal of this study is to examine the neurological outcome after endoscopic coronary artery bypass grafting (Endo-CABG). Endo-CABG is a minimal invasive cardiac procedure based on the conventional coronary artery bypass grafting (CABG) procedure.

Study design and study tests:

This study will be a single-centre prospective cohort study. The goal of the study is to assess the neurological outcome after endoscopic coronary artery bypass grafting (Endo-CABG). Three study groups will be included (described in section study groups), which will be tested for POCD, CVA and delirium.

Secondary outcomes in this research are quality of life of the patient (EQ-5D-5L), Fear and depression outcomes (VVO; CES-D), and assessment of demographic and peri-operative predictors of poor neurological outcome after endo-CABG.

Study tests:

Baseline tests will be performed in both intervention groups (Endo-CABG and PCI) and the healthy control group.

In the intervention groups the baseline preoperative tests will include:

* Baseline neurocognitive status: mini mental test
* Baseline EQ-5D: Quality of life
* Baseline fear and depression state (VVO; CES-D)
* Preoperative clinical neurological investigation
* Baseline POCD status (Rey auditory verbal learning test,Trailmaking A & B, Grooved pegboard test, Digit span test, Digit symbol-coding test)

For the healthy volunteers the same baseline tests will be performed, with exception of the neurological clinical evaluation.

Postoperative tests in the intervention groups will include:

* Postoperative neurologic clinical evaluation (CT scan if CVA suspected), CAM-ICU): these tests will be performed at the ICU or ward
* 3 months after surgery: EQ-5d (quality of life), Fear and depression, POCD follow-up (Rey auditory verbal learning test, Trailmaking A & B, Grooved pegboard test, Digit span test, Digit symbol-coding test)

For the healthy volunteers, the following tests will be performed 3 months after baseline testing:

* EQ-5d: quality of life
* Stroke follow-up
* Fear and depression
* POCD status (Rey auditory verbal learning test,Trailmaking A & B, Grooved pegboard test, Digit span test, Digit symbol-coding test)

Statistical analysis:

In this study POCD is defined as a decline in score between baseline and follow-up neurophysiological test, which should be higher than the natural variation. In this setting the natural learning effect will also be taken into account. To perform statistical analysis for POCD testing, Z-scores (or reliable change index (RCI)) will be used. The Z-score is a unit which indicates how the difference between the baseline score and the follow-up test behaves compared to the mean scores of the control group.

Thus, the individual RCI scores will be calculated as follows:

* For each patient, the baseline score from each test will be subtracted from the follow-up score, giving Δx. The same will be done in the control group, giving Δxc. The mean change on that test in the control group will then be subtracted from Δx to eliminate practice effects.
* This result will then be divided by the standard deviation of Δxc to eliminate the effect of natural variation in test performance. This is called a Z-score.

The RCI is the sum of the Z-scores of all tests.

We defined POCD in an individual patient as an RCI equal to or less than -1.645 (significance level 5%), or Z-score equal to or less than -1.645 in at least two different tests.

The group RCI scores will be compared using ANOVA or Kruskall-Wallis.

The quality of life will be tested using a mann-whitney U test at significance level 5%.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18
* Elective Endo-CABG procedure (group 1)
* Elective PCI procedure (group 2)
* Elective healthy volunteer

Exclusion Criteria:

* Medical history of:
* Postoperative cognitive dysfunction, delirium or cerebrovascular accident
* symptomatic carotid artery disease
* Dementia
* Renal dysfunction: glomular filtration rate (GFR) < 30 ml/min
* Hepatic dysfunction: serum glutamic-oxaloacetic transaminase (SGOT)/ aspartate aminotransferase (AST), or serum glutamic-pyruvic transaminase (SGPT)/ alanine aminotransferase (ALT), more than three timer higher than normal limits
* History of medication and alcohol abuse
* Language barrier or incapability to communicate
* Physical condition making participation impossible
* Participation in other clinical trials of a drug or medical instrument
* Surgical revision or intra-operative major cardial event (Endo-CABG group)
* Conversion to cardiac surgery or intra-operative major event (PCI group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be divided into three groups. The first group will be the Endo-CABG group which consist of the patients who undergo minimal invasive coronary artery bypass grafting.
  The second group consists of patients who will get an elective PCI intervention. this is a comparative group which is included to check whether the assessed prevalences in the Endo-CABG group are not related to underlying cardiac anomalies or to other cardiac intervention procedures.
  The third group consists of healthy volunteers. This control group will be included to eliminate natural variation in neurophysiological testing and to exclude the learning effect which can occur when repeated neurophysiological testing is performed.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of postoperative cognitive dysfunction | 3 months after intervention
  percentage of total study population
Prevalence of delirium | 3 months after intervention
  percentage of total study population
Prevalence of cerebrovascular accident | 3 months after intervention
  percentage of total study population

SECONDARY OUTCOMES:
Quality of life of the patient | 3 months after intervention
  assessment with the EQ-5D questionnaire
assessment of predictors of poor neurological outcome after minimal invasive coronary artery bypass grafting | 3 months after intervention
  assessment of which demographic and peri-operative variables are associated with poor neurological outcome after minimal invasive coronary
Incidence of depression after minimal invasive coronary artery bypass grafting | 3 months after intervention
  assessment with the CES-D questionnaire
Incidence of fear after minimal invasive coronary artery bypass grafting | 3 months after intervention
  assessment with the Surgical Fear Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Björn Stessel, MD, PhD, Principal Investigator — bjornstessel@hotmail.com
Locations (2):
- Belgium (2):
  - Jessa Hospital, Hasselt, Limburg
  - Jessaziekenhuis Hasselt, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Likosky DS, Nugent WC, Ross CS; Northern New England Cardiovascular Disease Study Group. Improving outcomes of cardiac surgery through cooperative efforts: the northern new England experience. Semin Cardiothorac Vasc Anesth. 2005 Jun;9(2):119-21. doi: 10.1177/108925320500900203. PMID 15920635
- [Background] GILMAN S. CEREBRAL DISORDERS AFTER OPEN-HEART OPERATIONS. N Engl J Med. 1965 Mar 11;272:489-98. doi: 10.1056/NEJM196503112721001. No abstract available. PMID 14250198
- [Background] Furlan AJ, Sila CA, Chimowitz MI, Jones SC. Neurologic complications related to cardiac surgery. Neurol Clin. 1992 Feb;10(1):145-66. PMID 1557000
- [Background] Jensen BO, Hughes P, Rasmussen LS, Pedersen PU, Steinbruchel DA. Health-related quality of life following off-pump versus on-pump coronary artery bypass grafting in elderly moderate to high-risk patients: a randomized trial. Eur J Cardiothorac Surg. 2006 Aug;30(2):294-9. doi: 10.1016/j.ejcts.2006.04.015. Epub 2006 Jul 7. PMID 16829089
- [Background] Newman MF, Grocott HP, Mathew JP, White WD, Landolfo K, Reves JG, Laskowitz DT, Mark DB, Blumenthal JA; Neurologic Outcome Research Group and the Cardiothoracic Anesthesia Research Endeavors (CARE) Investigators of the Duke Heart Center. Report of the substudy assessing the impact of neurocognitive function on quality of life 5 years after cardiac surgery. Stroke. 2001 Dec 1;32(12):2874-81. doi: 10.1161/hs1201.099803. PMID 11739990
- [Background] Newman MF. Open heart surgery and cognitive decline. Cleve Clin J Med. 2007 Feb;74 Suppl 1:S52-5. doi: 10.3949/ccjm.74.suppl_1.s52. No abstract available. PMID 17455545
- [Background] Ottens TH, Dieleman JM, Sauer AM, Peelen LM, Nierich AP, de Groot WJ, Nathoe HM, Buijsrogge MP, Kalkman CJ, van Dijk D; DExamethasone for Cardiac Surgery (DECS) Study Group. Effects of dexamethasone on cognitive decline after cardiac surgery: a randomized clinical trial. Anesthesiology. 2014 Sep;121(3):492-500. doi: 10.1097/ALN.0000000000000336. PMID 25225745
- [Background] Modi P, Chitwood WR Jr. Retrograde femoral arterial perfusion and stroke risk during minimally invasive mitral valve surgery: is there cause for concern? Ann Cardiothorac Surg. 2013 Nov;2(6):E1. doi: 10.3978/j.issn.2225-319X.2013.11.13. PMID 24350000
- [Derived] Stessel B, Nijs K, Pelckmans C, Vandenbrande J, Ory JP, Yilmaz A, Starinieri P, Van Tornout M, De Klippel N, Dendale P. Neurological outcome after minimally invasive coronary artery bypass surgery (NOMICS): An observational prospective cohort study. PLoS One. 2020 Dec 23;15(12):e0242519. doi: 10.1371/journal.pone.0242519. eCollection 2020. PMID 33362277
- [Derived] Nijs K, Vandenbrande J, Vaqueriza F, Ory JP, Yilmaz A, Starinieri P, Dubois J, Jamaer L, Arijs I, Stessel B. Neurological outcome after minimal invasive coronary artery surgery (NOMICS): protocol for an observational prospective cohort study. BMJ Open. 2017 Oct 6;7(10):e017823. doi: 10.1136/bmjopen-2017-017823. PMID 28988183